CLINICAL TRIAL: NCT04708392
Title: Stimulation Change Effects on Quantitative Sensory Testing in Neuromodulation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Burst 682552
Record Dates: First submitted 2020-07-07; First posted 2021-01-14 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tonic spinal cord stimulation (Experimental): Patients are programmed with tonic (continuous) spinal cord stimulation for a period of four weeks.
  Interventions: Device: Spinal Cord Stimulator
- Burst spinal cord stimulation (Experimental): Patients are programmed with burst (intermittent) spinal cord stimulation for a period of four weeks.
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — A spinal cord stimulator is a surgically implanted device that delivers an electrical signal to a patient's spinal cord to reduce the perception of pain

SUMMARY:
This study is designed to evaluate the effectiveness of two types of spinal cord stimulation programming types, in comparison to each other as well as patient baseline data.

DETAILED DESCRIPTION:
In this study patients have been implanted with an Abbott spinal cord stimulator capable of delivering both tonic (continuous) stimulation as well as Burst (intermittent) stimulation. Patients are programmed to be in both stimulation modes for a study period of 4 weeks, after which their pain symptoms are evaluated on a variety of surveys: McGill Pain Questionnaire (MPQ), Oswestry Disability Index (ODI), Beck Depression Inventory (BDI), Pain Catastrophizing Scale (PCS), Epworth Sleepiness Scale (ESS), Insomnia Severity Index (ISI), Numerical Rating Scale (NRS) and Global Improvement. They also undergo Quantitative Sensory Testing (QST), where thermal, mechanical, vibration and pressure stimuli are applied to the patient and detection limits are documented.

ELIGIBILITY:
Inclusion Criteria:

1. Albany Medical Center neurosurgery patients with chronic leg and/or back pain, that have, or are going to have, spinal cord stimulator implantation.
2. Patients are >/= 18 years old at the time of enrollment.
3. Patients must be: fluent in English; mentally competent; able to read and answer questionnaires; complete pain assessments; and give informed consent.

Exclusion Criteria:

1. Patients less than 18 years old.
2. Patients unable or unwilling to: read and answer questionnaires; complete pain assessments; and give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-29 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Quantitative Stimulus Testing (QST)-Thermal | Change from baseline to 4 weeks
  Thermal stimulus testing - thermal stimulation system is used to record hot and cold sensation and pain thresholds.

SECONDARY OUTCOMES:
McGill Pain Questionnaire (MPQ) | Change from baseline to 4 weeks
  This outcome measurement tool contains 15 descriptive words (11 sensory and 4 affective) used by subjects to describe their pain. Total number of words chosen is documented
Oswestry Disability Index (ODI) | Change from baseline to 4 weeks
  This measurement tool assesses functional outcome for 10 conditions in subjects with chronic pain. Patients select a statement for each condition that most closely resembles their own situation. Each statement has a score of 0-5, depending on the severity of the particular disability. Raw scores are calculated into a disability percentage.
Beck's Depression Inventory (BDI) | Change from baseline to 4 weeks
  This is a 21 section multiple-choice self-report survey. Patients select a statement in each section that most closely resembles their own situation. Each statement has a score of 0-3, depending on the severity of the depressive content. Raw scores are tallied.
Pain Catastrophizing Scale (PCS) | Change from baseline to 4 weeks
  This is a 13 question survey. It is used to assess the degree to which patients ruminate on, magnify, and/or amplify their pain symptoms. Patients rate on a scale of 0-4 (never - all the time) how often they have each of the thoughts listed. Raw scores are tallied
Numerical Rating Scale (NRS) | Change from baseline to 4 weeks
  Patients rate, on a scale of 0-10, their pain at it's least, most, and average over the past week. They also rate their pain "right now" as well as their perception of Global Improvement.
Epworth Sleepiness Scale (ESS) | Change from baseline to 4 weeks
  This survey is used to assess the 'daytime sleepiness' of patients. Patients rate the likelihood of falling asleep during several daytime scenarios, on a scale of 0-3 (never - very likely). Raw scores are tallied.
Insomnia Severity Index (ISI) | Change from baseline to 4 weeks
  This survey is designed to assess the nature, severity, and impact of insomnia in adults. Patients are asked to rate on a scale of 0-4 (no problem - very much a problem) how much of a problem they have with several sleep conditions. Raw scores are tallied.
Quantitative Stimulus Testing (QST)-Sensitivity | Change from baseline to 4 weeks
  Von Frey fibers are used to determine tactile sensitivity.
Quantitative Stimulus Testing (QST)-Pressure | Change from baseline to 4 weeks
  An algometer is used to measure pain related to pressure.
Quantitative Stimulus Testing (QST)-Vibration | Change from baseline to 4 weeks
  A tuning fork is used to measure sensitivity to vibration.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Pilitsis, MD, PhD, Principal Investigator — AMC Department of Neurosurgery
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Deer T, Slavin KV, Amirdelfan K, North RB, Burton AW, Yearwood TL, Tavel E, Staats P, Falowski S, Pope J, Justiz R, Fabi AY, Taghva A, Paicius R, Houden T, Wilson D. Success Using Neuromodulation With BURST (SUNBURST) Study: Results From a Prospective, Randomized Controlled Trial Using a Novel Burst Waveform. Neuromodulation. 2018 Jan;21(1):56-66. doi: 10.1111/ner.12698. Epub 2017 Sep 29. PMID 28961366
- [Background] Hou S, Kemp K, Grabois M. A Systematic Evaluation of Burst Spinal Cord Stimulation for Chronic Back and Limb Pain. Neuromodulation. 2016 Jun;19(4):398-405. doi: 10.1111/ner.12440. Epub 2016 May 3. PMID 27139915
- [Background] De Ridder D, Plazier M, Kamerling N, Menovsky T, Vanneste S. Burst spinal cord stimulation for limb and back pain. World Neurosurg. 2013 Nov;80(5):642-649.e1. doi: 10.1016/j.wneu.2013.01.040. Epub 2013 Jan 12. PMID 23321375